CLINICAL TRIAL: NCT00607386
Title: A Multi-Center, Open-Label Study Evaluating Safety and Clinical Outcomes in Hunter Syndrome Patients 5 Years of Age and Younger Receiving Idursulfase Enzyme Replacement Therapy
Brief Title: Safety and Clinical Outcomes in Hunter Syndrome Patients 5 Years of Age and Younger Receiving Idursulfase Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Covance (Industry); PharmaNet (Industry); PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-ELA-038; 2007-006044-22 (EudraCT Number)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hunter Syndrome; Mucopolysaccharidosis II; MPS II
Keywords: Hunter syndrome; hunters syndrome; hunter's syndrome; hunter disease; hunters disease; hunter's disease; MPS II; MPSII; MPS2; MPS 2; mucopolysaccharides; lysosomal storage disease; lysosomal storage disorder; chronic ear infection; enlarged adenoids; mps symptoms; mps diagnosis; mps ii therapy; MPS II treatment; ert treatment; elaprase; idursulfase; iduronate sulfatase; iduronate 2 sulfatase; enzyme replacement therapy; hunter syndrome treatment; hunter's syndrome treatment; hunter syndrome therapy; hunter's disease treatment; mps society
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases | interventions — idursulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idursulfase (Other): Open-label treatment with idursulfase
  Interventions: Biological: Idursulfase

INTERVENTIONS:
Biological: Idursulfase — Solution for intravenous infusion, 0.5 mg/kg weekly
  Other Names: Elaprase

SUMMARY:
The objective of this study is to determine the safety of once weekly dosing of idursulfase 0.5 mg/kg administered by intravenous (IV) infusion for male Hunter syndrome patients ≤ 5 years old.

DETAILED DESCRIPTION:
This study will provide a basis for evaluating the safety of idursulfase administered to Hunter syndrome patients who are ≤ 5 years old. Additionally, this study will provide a basis for evaluating the idursulfase single- and repeated-dose pharmacokinetic profiles as well as the pharmacodynamic effect (as measured by urinary GAG excretion) in this pediatric population. Additional exploratory measures will include abdominal ultrasound measurements of liver and spleen volumes, assessments of growth with comparisons to normal population growth data, assessments of annualized growth velocity, assessments of routine developmental milestones using the Denver II, and assessments of clinical events, including the first occurrence of certain hearing-related events (e.g., hearing loss, otitis media), respiratory-related events (e.g., upper and lower respiratory infections), and specific surgical procedures (e.g., adenoidectomy, placement of PE tubes).

All patients in this open-label study will receive once-weekly infusions of idursulfase at a dose of 0.5 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of Hunter syndrome based upon biochemical criteria either documented in their medical history or established at Screening:

  1. A deficiency in iduronate-2-sulfatase (I2S) enzyme activity of ≤ 10 % of the lower limit of the normal range as measured in plasma, fibroblasts, or leukocytes (based on normal range of measuring laboratory)

     AND
  2. A normal enzyme activity level of one other sulfatase as measured in plasma, fibroblasts, or leukocytes (based on normal range of measuring laboratory).
* The patient is 5 years of age and under.
* The patient is male.
* The patient's parent(s), or patient's legal guardian must have voluntarily signed an Institutional Review Board approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient's parent(s), or the patient's legal guardian.

Exclusion Criteria:

* The patient has received treatment with another investigational therapy within 30 days prior to enrollment.
* The patient has clinically relevant medical condition(s) making implementation of the protocol difficult.
* The patient has previously received idursulfase.
* The patient has known hypersensitivity to any of the components of idursulfase.
* The patient has had a tracheostomy.

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2007-12-31 (Actual); Primary Completion 2011-07-08 (Actual); Study Completion 2011-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Hospital de Clinicas de Porto Alegre, Servico de Genetica Medica, Porto Alegre, Rio Grande do Sul, Brazil
- Instytut Pomnik Centrum Zdrowia Dziecka, Klinika Chorob Metaboliczynch, Endokrynologii i Diabetologii, Warsaw, Poland
- National Taiwan University Hospital, Dept. of Pediatrics and Medical Genetics, Taipei, Taiwan

REFERENCES:
- [Background] Muenzer J, Gucsavas-Calikoglu M, McCandless SE, Schuetz TJ, Kimura A. A phase I/II clinical trial of enzyme replacement therapy in mucopolysaccharidosis II (Hunter syndrome). Mol Genet Metab. 2007 Mar;90(3):329-37. doi: 10.1016/j.ymgme.2006.09.001. Epub 2006 Dec 20. PMID 17185020
- [Background] Muenzer J, Wraith JE, Beck M, Giugliani R, Harmatz P, Eng CM, Vellodi A, Martin R, Ramaswami U, Gucsavas-Calikoglu M, Vijayaraghavan S, Wendt S, Puga AC, Ulbrich B, Shinawi M, Cleary M, Piper D, Conway AM, Kimura A. A phase II/III clinical study of enzyme replacement therapy with idursulfase in mucopolysaccharidosis II (Hunter syndrome). Genet Med. 2006 Aug;8(8):465-73. doi: 10.1097/01.gim.0000232477.37660.fb. PMID 16912578
- [Result] Pano A, Barbier AJ, Bielefeld B, Whiteman DA, Amato DA. Immunogenicity of idursulfase and clinical outcomes in very young patients (16 months to 7.5 years) with mucopolysaccharidosis II (Hunter syndrome). Orphanet J Rare Dis. 2015 Apr 24;10:50. doi: 10.1186/s13023-015-0265-2. PMID 25902842

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Idursulfase
Started | 28
Completed | 27
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all enrolled participants who received at least one study dose (or any portion of a dose) of idursulfase.
Arm/Group | Idursulfase
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.0 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Baseline Normalized Urinary Glycosaminoglycan (GAG) Level [Mean (Standard Deviation); unit: microgram per milligram creatinine] | 738.3 (165.21)

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that did not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with AEs occurred after start of study treatment until 30 days after the last infusion of idursulfase, were reported.
Time Frame: From the start of study treatment until 30 days after the last infusion of idursulfase, up to 53 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Idursulfase
Number analyzed (Participants) | 28
participants
  Experienced at least one adverse event (AE) | 28
  Deaths | 0
  Discontinued due to an AE | 0
  Experienced at least one drug-related AE | 16
  Experienced at least one serious AE (SAE) | 13
  Experienced at least one severe AE | 2
  Experienced at least one infusion-related AE | 16

2. Secondary Outcome: Mean Change From Baseline to Week 53 in Normalized Urinary Glycosaminoglycan (GAG) Levels
Description: Analysis of urinary GAG levels was performed at baseline, Week 18, Week 36, and Week 53 as an assessment of the pharmacodynamic effects of Elaprase (idursulfase).
Time Frame: Baseline, Weeks 18, 36 and 53
Population: Safety population. In the categories listed below, 'N' signifies the number of participants evaluable for the timepoint.
Measure: Mean (Standard Deviation); unit: microgram/milligram creatinine
Arm/Group | Idursulfase
Number analyzed (Participants) | 28
microgram/milligram creatinine
  Baseline (N=28) | 738.3 (165.21)
  Change at Week 18 (N=27) | -368.0 (165.44)
  Change at Week 36 (N=27) | -400.3 (180.27)
  Change at Week 53 (N=27) | -402.4 (162.13)

3. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Maximum Observed Serum Concentration (Cmax)
Time Frame: Weeks 1 and 27
Population: Pharmacokinetic (PK) population was defined as all enrolled participants who had at least one serum concentration measurement available. In the categories listed below, "N" signifies the number of participants evaluable for the timepoint.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Idursulfase
Number analyzed (Participants) | 27
nanogram per milliliter
  Week 1 (N=27) | 1333 (817)
  Week 27 (N=19) | 1032 (590)

4. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Time of Maximum Observed Serum Concentration (Tmax)
Time Frame: Weeks 1 and 27
Population: PK population. In the categories listed below, "N" signifies the number of participants evaluable for the timepoint.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Idursulfase
Number analyzed (Participants) | 27
minutes
  Week 1 (N=27) | 163 (28)
  Week 27 (N=19) | 167 (32)

5. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Area Under the Serum Concentration-Time Curve From Time 0 to the Final Time Point With a Concentration of at Least Lower Limit of Quantitation (AUClast)
Time Frame: Weeks 1 and 27
Population: PK population. In the categories listed below, "N" signifies the number of participants evaluable for the timepoint.
Measure: Mean (Standard Deviation); unit: minute*nanogram per milliliter
Arm/Group | Idursulfase
Number analyzed (Participants) | 27
minute*nanogram per milliliter
  Week 1 (N=27) | 196526 (71779)
  Week 27 (N=19) | 174869 (109118)

6. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUCinf)
Time Frame: Weeks 1 and 27
Population: PK population with evaluable participants for this endpoint. In the categories listed below, "N" signifies the number of participants evaluable for the timepoint.
Measure: Mean (Standard Deviation); unit: minute*nanogram per milliliter
Arm/Group | Idursulfase
Number analyzed (Participants) | 26
minute*nanogram per milliliter
  Week 1 (N=26) | 224343 (76944)
  Week 27 (N=18) | 201130 (117575)

7. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Elimination Half-Life (t1/2)
Description: t1/2 refers to the elimination of the drug. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase of elimination. It is expressed in minutes and derived from the terminal slope of the concentration versus time curve.
Time Frame: Weeks 1 and 27
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Idursulfase
Number analyzed (Participants) | 26
minutes
  Week 1 (N=26) | 160 (69)
  Week 27 (N=18) | 109 (43)

8. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Mean Residence Time From Time 0 to Infinity (MRTinf)
Description: MRTinf is an average duration of the drug in the body from time zero to infinity, and is expressed in minutes.
Time Frame: Weeks 1 and 27
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Idursulfase
Number analyzed (Participants) | 26
minutes
  Week 1 (N=26) | 153 (96)
  Week 27 (N=18) | 127 (23)

9. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Clearance (CL)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Weeks 1 and 27
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliter/minute/kilogram
Arm/Group | Idursulfase
Number analyzed (Participants) | 26
milliliter/minute/kilogram
  Week 1 (N=26) | 2.4 (0.7)
  Week 27 (N=18) | 4.7 (5.0)

10. Secondary Outcome: Single- and Repeat-Dose Pharmacokinetics - Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steadystate.
Time Frame: Weeks 1 and 27
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliter per kilogram
Arm/Group | Idursulfase
Number analyzed (Participants) | 26
milliliter per kilogram
  Week 1 (N=26) | 394 (423)
  Week 27 (N=18) | 551 (528)

ADVERSE EVENTS:
Time Frame: From the start of study treatment until 30 days after the last infusion of idursulfase, up to 53 weeks
Arm/Group | Idursulfase
Serious Adverse Events (participants affected / at risk) | 13/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idursulfase (N=28)
Bronchopneumonia (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 3 (6)
Catheter site haematoma (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Atonic seizures (Nervous system disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.57% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idursulfase (N=28)
Upper respiratory tract infection (Infections and infestations) | 18 (42)
Respiratory tract infection (Infections and infestations) | 12 (36)
Rhinitis (Infections and infestations) | 11 (20)
Viral upper respiratory tract infection (Infections and infestations) | 9 (17)
Otitis media acute (Infections and infestations) | 7 (10)
Pharyngitis (Infections and infestations) | 7 (18)
Gastroenteritis (Infections and infestations) | 6 (7)
Upper respiratory tract infection bacterial (Infections and infestations) | 6 (13)
Pneumonia (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 5 (6)
Bronchitis (Infections and infestations) | 4 (4)
Bronchopneumonia (Infections and infestations) | 3 (4)
Otitis media (Infections and infestations) | 2 (3)
Gastrointestinal infection (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 3 (5)
Viral infection (Infections and infestations) | 3 (4)
Viral pharyngitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Herpes virus infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Laryngitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Body tinea (Infections and infestations) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lice infestation (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (2)
Varicella (Infections and infestations) | 1 (1)
Viral diarrhoea (Infections and infestations) | 1 (2)
Pyrexia (General disorders) | 25 (59)
Fatigue (General disorders) | 2 (2)
Catheter site haematoma (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Malaise (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (45)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (11)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (7)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Heat rash (Skin and subcutaneous tissue disorders) | 2 (4)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (12)
Diarrhoea (Gastrointestinal disorders) | 7 (35)
Constipation (Gastrointestinal disorders) | 2 (3)
Dental caries (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Anal fissure (Gastrointestinal disorders) | 1 (2)
Faeces hard (Gastrointestinal disorders) | 1 (2)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Pruritus ani (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 4 (4)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (2)
Conductive deafness (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Agitation (Psychiatric disorders) | 4 (5)
Sleep disorder (Psychiatric disorders) | 3 (3)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Crying (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Learning disorder (Psychiatric disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 4 (4)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1)
Right ventricular hypertrophy (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Lymphocyte morphology abnormal (Investigations) | 1 (1)
Monocyte count decreased (Investigations) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Atonic seizures (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hyperaemia (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Lordosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Hypermetropia (Eye disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1)
Hip dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.